CLINICAL TRIAL: NCT00584870
Title: PHASE II RANDOMIZED, DOUBLE-BLIND, PLACEBO-AND ACTIVE CONTROLLED, MULTICENTER, PARALLEL GROUP PROOF OF CONCEPT STUDY OF THE ANALGESIC EFFECTS OF RN624 IN ADULT PATIENTS WITH CHRONIC LOW BACK PAIN
Brief Title: RN624 In Adult Patients With Chronic Low Back Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A4091004; CLBP POC (Other: Alias Study Number)
Record Dates: First submitted 2007-12-21; First posted 2008-01-02 (Estimated); Results first posted 2021-06-16 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2021-06

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Naproxen; tanezumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Naproxen (Active Comparator)
  Interventions: Drug: Naproxen
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- RN624 (Experimental)
  Interventions: Drug: PF-04383119 (RN624)

INTERVENTIONS:
Drug: Naproxen — Oral naproxen 500 mg twice daily for Weeks 1-12.
  Arms: Naproxen
Drug: Placebo — Single IV infusion of placebo on Day 1 and placebo for naproxen twice daily for Weeks 1-12.
  Arms: Placebo
Drug: PF-04383119 (RN624) — Single IV infusion of 200 micrograms/kg RN624 on Day 1
  Arms: RN624

SUMMARY:
The primary objective of this study is to evaluate the analgesic efficacy of RN624 compared with placebo and compared with naproxen in the treatment of adult patients with chronic low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Male or female of any race, >18 years of age and have BMI ≤39 kg/m2
* Present with duration of chronic low back pain of ≥3 months requiring regular use of analgesic medication (>4 days per week for the past month)
* Primary location of low back pain is between the 12th thoracic vertebra and the lower gluteal folds, with or without radiation into the posterior thigh, classified as Category 1 or 2 according to the classification of the Quebec Task Force in Spinal Disorders
* Must have a score of ≥4 for Low Back Pain Intensity (NRS) while on current treatment at Screening, and completes at least 4 daily pain diaries during the 5 days prior to Randomization, with an average Low Back Pain Intensity (NRS) score of ≥4

Exclusion Criteria:

* Back pain due to visceral disorder (i.e. endometriosis) or Back pain due to recent major trauma (i.e. vertebral fracture, post-traumatic spondylolisthesis)
* History of lumbosacral radiculopathy, spinal stenosis associated with neurological impairment, or neurogenic claudication
* Osteoporotic compression fracture within the last 6 months
* Known history of: Rheumatoid arthritis; Seronegative spondyloarthropathy (i.e., ankylosing spondylitis, psoriatic arthritis, reactive arthritis, inflammatory bowel disease-related arthropathy); Paget's disease of spine, pelvis or femur; Fibromyalgia; Tumors or infections of the spinal cord
* Patients receiving acetaminophen only to manage their chronic low back pain
* Any uncontrolled or untreated chronic disease

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2007-07-05 (Actual); Primary Completion 2008-09-02 (Actual); Study Completion 2008-09-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (38):
- United States (38):
  - Pinnacle Research Group LLC, Anniston, Alabama
  - Radiant Research, Birmingham, Alabama
  - Radiant Research - Phoenix Southeast, Chandler, Arizona
  - Radiant Research, Scottsdale, Arizona
  - Advanced Clinical Research Institute, Anaheim, California
  - University of California San Diego, San Diego, California
  - Doctors Medical Center of Walton County, DeFuniak Springs, Florida
  - SJS Clinical Research, Inc., Destin, Florida
  - Adult Medicine Specialists, Longwood, Florida
  - Genesis Research International, Longwood, Florida
  - Collier Neurologic Specialists, Naples, Florida
  - Cotton-O'Neil Clinical Research, Topeka, Kansas
  - Cotton-O'Neil Clinic, Topeka, Kansas
  - Heartland Research Associates, Wichita, Kansas
  - Northeast Medical Research Associates, Inc, North Dartmouth, Massachusetts
  - Clinical Pharmacology Study Group, Worcester, Massachusetts
  - Spence Medical Research, Picayune, Mississippi
  - Radiant Research, Inc., St Louis, Missouri
  - Quality Clinical Research, Inc., Omaha, Nebraska
  - The Medical Research Network, LLC, New York, New York
  - North State Clinical Research, PLLC, Lenoir, North Carolina
  - Wake Internal Medicine Consultants, Inc., Raleigh, North Carolina
  - Wake Research Associates, Raleigh, North Carolina
  - Summit Research Network (Oregon), Inc., Portland, Oregon
  - Allegheny Pain Management, Altoona, Pennsylvania
  - New England Center for Clinical Research, Cranston, Rhode Island
  - Partners in Clinical Research, Cumberland, Rhode Island
  - Omega Medical Research, Warwick, Rhode Island
  - Radiant Research, Greer, South Carolina
  - Advanced Therapeutics, Inc., Johnson City, Tennessee
  - Johnson City Internal Medicine, Johnson City, Tennessee
  - DiscoveResearch, Incorporated, Bryan, Texas
  - Advances In Health, Inc., Houston, Texas
  - Centex Research, Nassau Bay, Texas
  - Immediate Medical Care, Nassau Bay, Texas
  - Radiant Research San Antonio, San Antonio, Texas
  - Independence Family Medicine, Virginia Beach, Virginia
  - Summit Research Network (Seattle) LLC, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4091004&StudyName=RN624%20In%20Adult%20Patients%20With%20Chronic%20Low%20Back%20Pain

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants underwent a 5-day initial pain assessment period prior to study treatment.
Groups:
- Tanezumab: Single intravenous infusion of tanezumab (RN624 or PF-04383119) 200 microgram per kilogram (mcg/kg) at Baseline (Day 1) along with placebo matched to naproxen tablet orally twice daily up to Week 12.
- Naproxen: Single intravenous infusion of placebo matched to tanezumab (RN624 or PF-04383119) at Baseline (Day 1) along with naproxen 500 milligram (mg) tablet orally twice daily up to Week 12.
- Placebo: Single intravenous infusion of placebo matched to tanezumab (RN624 or PF-04383119) at Baseline (Day 1) along with placebo matched to naproxen tablet orally twice daily up to Week 12.
Period: Overall Study
Arm/Group | Tanezumab | Naproxen | Placebo
Started | 88 | 89 | 43
Treated | 88 | 88 | 41
Completed | 59 | 64 | 25
Not Completed | 29 | 25 | 18
Not completed — Adverse Event | 4 | 3 | 2
Not completed — Lost to Follow-up | 4 | 1 | 1
Not completed — Lack of Efficacy | 7 | 14 | 8
Not completed — Withdrawal by Subject | 10 | 5 | 3
Not completed — Protocol Violation | 1 | 1 | 2
Not completed — Did not met entrance criteria | 1 | 0 | 0
Not completed — Other | 2 | 0 | 0
Not completed — Randomized but not treated | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Population: Intent to treat (ITT) population included all randomized participants who received the Day 1 intravenous infusion (either tanezumab or placebo infusion).
Groups:
- Total: Total of all reporting groups
Arm/Group | Tanezumab | Naproxen | Placebo | Total
Number analyzed (Participants) | 88 | 88 | 41 | 217
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.5 (14.7) | 52.1 (14.8) | 52.2 (15) | 51.1 (14.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 42 | 23 | 118
  Male | 35 | 46 | 18 | 99

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Daily Average Low Back Pain Intensity (LBPI) Score at Week 6
Description: Daily average low back pain was assessed on an 11-point numeric rating scale (NRS). Participants described their average low back pain during the past 24 hours on a scale ranging from 0 (no pain) to 10 (worst possible pain). Baseline value was calculated as mean of the scores over 5-day prior to randomization (initial pain assessment period). Post-baseline weekly scores were calculated based on the mean of the scores over the 7 days prior to and including the day at the end of the corresponding week.
Time Frame: Baseline, Week 6
Population: ITT population included all randomized participants who received the Day 1 intravenous infusion (either tanezumab or placebo infusion). Here 'number analyzed' signifies participants who were evaluable for this measure at given time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab | Naproxen | Placebo
Number analyzed (Participants) | 88 | 88 | 41
units on a scale
  Baseline | 6.48 (1.42) | 6.65 (1.44) | 6.67 (1.44)
  Change at Week 6: number analyzed (Participants) | 67 | 76 | 33
  Change at Week 6 | -3.58 (1.87) | -2.69 (1.98) | -2.16 (2.24)
Statistical Analysis 1: Comparison: Tanezumab vs Placebo; LS mean difference was estimated from the repeated measures model with baseline, center, treatment, week and treatment-by-week interaction as fixed main effects and participant as random effect; Test type: Superiority or Other; p = 0.001, Repeated Measures Model — p-value was based on repeated measures model from pairwise comparisons, and statistical test was 1-sided with 0.1 significance level; Least squares (LS) Mean Difference = -1.17, 80% CI 2-sided [-1.67 to -0.67], Standard Error of Mean 0.39

2. Secondary Outcome: Change From Baseline in Daily Average Low Back Pain Intensity (LBPI) Score at Week 1, 2, 4, 8 and 12
Description: Daily average low back pain was assessed on an 11-point numeric rating scale (NRS). Participants described their average low back pain during the past 24 hours on a scale ranging from 0 (no pain) to 10 (worst possible pain), with lower scores indicating less pain. Baseline value was calculated as mean of the scores over 5-day prior to randomization (initial pain assessment period). Post-baseline weekly scores were calculated based on the mean of the scores over the 7 days prior to and including the day at the end of the corresponding week.
Time Frame: Baseline, Week 1, 2, 4, 8, 12
Population: ITT population included all randomized participants who received the Day 1 intravenous infusion (either tanezumab or placebo infusion). Here "overall number of participants analyzed" signifies those participants who were evaluable for this outcome measure and 'number analyzed' signifies those participants who were evaluable for this measure at given time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab | Naproxen | Placebo
Number analyzed (Participants) | 88 | 87 | 40
units on a scale
  Change at Week 1 | -2.41 (1.69) | -2.18 (1.81) | -1.34 (1.52)
  Change at Week 2: number analyzed (Participants) | 83 | 87 | 39
  Change at Week 2 | -2.25 (2.04) | -2.40 (1.83) | -1.92 (1.87)
  Change at Week 4: number analyzed (Participants) | 74 | 79 | 37
  Change at Week 4 | -3.39 (1.83) | -2.57 (1.86) | -2.23 (2.07)
  Change at Week 8: number analyzed (Participants) | 64 | 71 | 31
  Change at Week 8 | -3.74 (1.88) | -2.79 (2.06) | -2.48 (2.09)
  Change at Week 12: number analyzed (Participants) | 58 | 65 | 26
  Change at Week 12 | -3.45 (2.08) | -2.88 (2.24) | -2.68 (2.40)

3. Secondary Outcome: Change From Baseline in Average Low Back Pain Intensity (LBPI) Score Over Weeks 1 to 4, 1 to 8, 1 to 12, 5 to 8, and 5 to 12
Description: Daily average low back pain was assessed on an 11-point numeric rating scale (NRS). Participants described their average low back pain during the past 24 hours on a scale ranging from 0 (no pain) to 10 (worst possible pain), with lower scores indicating less pain. Baseline value was calculated as mean of the scores over 5-day prior to randomization (initial pain assessment period). Post-baseline weekly scores were calculated based on the mean of the scores over the 7 days prior to and including the day at the end of the corresponding week. Change from baseline was calculated as the average of each specified week interval (Week 1 to 4, 1 to 8, 1 to 12, 5 to 8, 5 to 12) values minus the baseline value.
Time Frame: Baseline, Weeks 1 to 4, 1 to 8, 1 to 12, 5 to 8, 5 to 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab | Naproxen | Placebo
Number analyzed (Participants) | 88 | 87 | 41
units on a scale
  Change over Weeks 1 to 4 | -2.59 (1.75) | -2.35 (1.73) | -1.83 (1.71)
  Change over Weeks 1 to 8 | -2.86 (1.81) | -2.47 (1.75) | -1.97 (1.80)
  Change over Weeks 1 to 12 | -2.92 (1.85) | -2.52 (1.80) | -2.06 (1.84)
  Change over Weeks 5 to 8: number analyzed (Participants) | 69 | 78 | 34
  Change over Weeks 5 to 8 | -3.56 (1.91) | -2.66 (1.89) | -2.38 (2.07)
  Change over Weeks 5 to 12: number analyzed (Participants) | 69 | 78 | 34
  Change over Weeks 5 to 12 | -3.48 (1.94) | -2.68 (1.94) | -2.46 (2.07)

4. Secondary Outcome: Change From Baseline in Modified Brief Pain Inventory-short Form (mBPI-sf) Scores for Worst Pain and Average Pain at Week 1, 2, 4, 6, 8 and 12
Description: The mBPI-sf was a self-administered questionnaire used to assess the severity of pain and the impact of pain on daily functions during the 24-hour period prior to evaluation. It consisted of 5 questions. Questions (Q) 1-4 assessed the magnitude of pain (Q1 for worst pain, Q2 for least pain, Q3 for average pain, Q4 for pain right now) on an 11-point NRS ranging from 0 (no pain) to 10 (pain as bad as you can imagine), with lower scores indicating less pain. Question 5 consisted of 7 sub-items (A to G; general activity, mood, walking ability, normal work, relations with other people, sleep, enjoyment of life) which measured the level of interference of pain on daily functions. Each sub-item was assessed on an 11-point NRS ranging from 0 (does not interfere) to 10 (completely interferes). Results are reported for worst and average pain score, each ranging from 0 (no pain) to 10 (pain as bad as you can imagine), with lower scores indicating less pain.
Time Frame: Baseline, Week 1, 2, 4, 6, 8, 12
Population: ITT population included all randomized participants who received the Day 1 intravenous infusion (either tanezumab or placebo infusion). Here 'number analyzed' signifies those participants who were evaluable for this measure at given time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab | Naproxen | Placebo
Number analyzed (Participants) | 88 | 88 | 41
units on a scale
  Baseline: Worst Pain | 6.89 (1.69) | 7.02 (1.74) | 7.29 (1.65)
  Baseline: Average Pain | 5.99 (1.43) | 6.18 (1.42) | 6.54 (1.64)
  Change at Week 1: Worst Pain: number analyzed (Participants) | 78 | 83 | 41
  Change at Week 1: Worst Pain | -2.54 (2.33) | -2.40 (2.02) | -1.88 (2.38)
  Change at Week 1: Average Pain: number analyzed (Participants) | 78 | 83 | 41
  Change at Week 1: Average Pain | -2.09 (2.07) | -2.02 (1.77) | -1.46 (1.95)
  Change at Week 2: Worst Pain: number analyzed (Participants) | 77 | 82 | 36
  Change at Week 2: Worst Pain | -2.21 (2.53) | -2.67 (2.24) | -2.28 (2.25)
  Change at Week 2: Average Pain: number analyzed (Participants) | 77 | 82 | 36
  Change at Week 2: Average Pain | -1.97 (2.01) | -2.20 (1.82) | -2.22 (2.22)
  Change at Week 4: Worst Pain: number analyzed (Participants) | 69 | 79 | 36
  Change at Week 4: Worst Pain | -3.54 (2.17) | -2.57 (2.29) | -2.47 (3.25)
  Change at Week 4: Average Pain: number analyzed (Participants) | 69 | 79 | 36
  Change at Week 4: Average Pain | -2.99 (1.91) | -2.37 (1.87) | -2.61 (2.56)
  Change at Week 6: Worst Pain: number analyzed (Participants) | 66 | 75 | 31
  Change at Week 6: Worst Pain | -3.67 (2.45) | -2.87 (2.34) | -2.29 (3.30)
  Change at Week 6: Average Pain: number analyzed (Participants) | 66 | 75 | 31
  Change at Week 6: Average Pain | -3.29 (1.85) | -2.45 (1.98) | -2.65 (2.39)
  Change at Week 8: Worst Pain: number analyzed (Participants) | 61 | 71 | 30
  Change at Week 8: Worst Pain | -3.85 (2.37) | -2.89 (2.56) | -2.90 (2.77)
  Change at Week 8: Average Pain: number analyzed (Participants) | 61 | 71 | 30
  Change at Week 8: Average Pain | -3.26 (1.89) | -2.44 (2.03) | -2.80 (2.30)
  Change at Week 12: Worst Pain: number analyzed (Participants) | 60 | 67 | 24
  Change at Week 12: Worst Pain | -3.40 (2.37) | -2.93 (2.66) | -2.83 (3.17)
  Change at Week 12: Average Pain: number analyzed (Participants) | 60 | 67 | 24
  Change at Week 12: Average Pain | -3.00 (1.92) | -2.45 (2.36) | -2.88 (2.47)

5. Secondary Outcome: Number of Participants With Average Low Back Pain Intensity (LBPI) Score of 2 or Less
Description: Daily average low back pain was assessed on an 11-point numeric rating scale (NRS). Participants described their average low back pain during the past 24 hours on a scale ranging from 0 (no pain) to 10 (worst possible pain), with lower scores indicating less pain. Weekly scores were calculated based on the mean of the scores over the 7 days prior to and including the day at the end of the corresponding week. Participants were classified as responders if average LBPI score was 2 or less, and as non-responders if average LBPI score was greater than (>) 2. Participants with average LBPI score of 2 or less were reported.
Time Frame: Week 1, 2, 4, 6, 8, 12
Population: ITT population included all randomized participants who received the Day 1 intravenous infusion (either tanezumab or placebo infusion). Last observation carried forward (LOCF) method was used to impute missing values.
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab | Naproxen | Placebo
Number analyzed (Participants) | 88 | 88 | 41
Participants
  Week 1 | 18 | 13 | 2
  Week 2 | 20 | 19 | 4
  Week 4 | 27 | 19 | 6
  Week 6 | 33 | 21 | 5
  Week 8 | 32 | 25 | 8
  Week 12 | 26 | 21 | 6

6. Secondary Outcome: Number of Participants With Cumulative Percent (%) Reduction From Baseline in Average Low Back Pain Intensity (LBPI) Score at Week 6
Description: Daily average low back pain was assessed on an 11-point numeric rating scale (NRS). Participants described their average low back pain during the past 24 hours on a scale ranging from 0 (no pain) to 10 (worst possible pain), with lower scores indicating less pain. Baseline value was calculated as mean of the scores over 5-day prior to randomization (initial pain assessment period). Post-baseline weekly scores were calculated based on the mean of the scores over the 7 days prior to and including the day at the end of the corresponding week. Number of participants with cumulative reduction (as percent) (greater than 0% ; >= 10, 20, 30, 40, 50, 60, 70, 80 and 90%; = 100 %) in Average LBPI score from Baseline at Week 6 were reported, participants (%) are reported more than once in categories specified.
Time Frame: Week 6
Population: ITT population included all randomized participants who received the Day 1 intravenous infusion (either tanezumab or placebo infusion). LOCF method was used to impute missing values.
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab | Naproxen | Placebo
Number analyzed (Participants) | 88 | 88 | 41
Participants
  Greater than 0% reduction | 79 | 77 | 34
  Greater than or equal to (>=)10% reduction | 75 | 72 | 29
  >=20% reduction | 68 | 64 | 21
  >=30% reduction | 65 | 50 | 13
  >=40% reduction | 58 | 41 | 12
  >=50% reduction | 50 | 30 | 8
  >=60% reduction | 40 | 26 | 7
  >=70% reduction | 25 | 16 | 5
  >=80% reduction | 16 | 9 | 3
  >=90% reduction | 10 | 5 | 1
  100% reduction | 6 | 3 | 0

7. Secondary Outcome: Number of Participants With at Least 30% and 50% Sustained Reduction From Baseline in Daily Average Low Back Pain Intensity (LBPI) Score
Description: Daily average low back pain was assessed on an 11-point numeric rating scale (NRS). Participants described their average low back pain during the past 24 hours on a scale ranging from 0 (no pain) to 10 (worst possible pain) with lower scores indicating less pain. Baseline value was calculated as mean of the scores over 5-day prior to randomization (initial pain assessment period). Post-baseline weekly scores were calculated based on the mean of the scores over the 7 days prior to and including the day at the end of the corresponding week. Participants with >=30% or >=50% reduction from baseline in daily average LBPI score that was maintained for a minimum duration of 4 consecutive days were reported.
Time Frame: Week 12
Population: ITT population included all randomized participants who received the Day 1 intravenous infusion (either tanezumab or placebo infusion). Here '"overall number of participants analyzed" signifies those participants who were evaluable for this outcome measure
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab | Naproxen | Placebo
Number analyzed (Participants) | 88 | 87 | 41
Participants
  >=30% reduction | 71 | 60 | 26
  >=50% reduction | 62 | 50 | 20

8. Secondary Outcome: Number of Participants With at Least 30% and 50% Reduction From Baseline in Daily Average Low Back Pain Intensity (LBPI) Score
Description: Daily average low back pain was assessed on an 11-point numeric rating scale (NRS). Participants described their average low back pain during the past 24 hours on a scale ranging from 0 (no pain) to 10 (worst possible pain), with lower scores indicating less pain. Baseline value was calculated as mean of the scores over 5-day prior to randomization (initial pain assessment period). Post-baseline weekly scores were calculated based on the mean of the scores over the 7 days prior to and including the day at the end of the corresponding week. Number of participants with >=30% and >=50% reduction from Baseline in daily average LBPI score were reported.
Time Frame: Weeks 1, 2, 4, 6, 8, 12
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab | Naproxen | Placebo
Number analyzed (Participants) | 88 | 88 | 41
Participants
  Week 1: >=30% reduction | 46 | 45 | 8
  Week 1: >=50% reduction | 28 | 26 | 5
  Week 2: >=30% reduction | 42 | 48 | 14
  Week 2: >=50% reduction | 28 | 31 | 7
  Week 4: >=30% reduction | 62 | 50 | 16
  Week 4: >=50% reduction | 43 | 28 | 10
  Week 6: >=30% reduction | 65 | 50 | 13
  Week 6: >=50% reduction | 50 | 30 | 8
  Week 8: >=30% reduction | 66 | 51 | 18
  Week 8: >=50% reduction | 49 | 33 | 9
  Week 12: >=30% reduction | 59 | 45 | 20
  Week 12: >=50% reduction | 43 | 30 | 12

9. Secondary Outcome: Time to Achieve at Least 30% and 50% Sustained Reduction From Baseline in Daily Average Low Back Pain Intensity (LBPI) Score
Description: Time to achieve >=30% or >=50% sustained reduction from baseline (i.e. reduction from baseline in daily average LBPI score that was maintained for a total of 4 consecutive days) was summarized using the Kaplan-Meier estimates of the median time to 30% and 50% response. Daily average low back pain was assessed on an 11-point numeric rating scale (NRS). Participants described their average low back pain during the past 24 hours on a scale ranging from 0 (no pain) to 10 (worst possible pain), with lower scores indicating less pain. Baseline value was calculated as mean of the scores over 5-day prior to randomization (initial pain assessment period). Post-baseline weekly scores were calculated based on the mean of the scores over the 7 days prior to and including the day at the end of the corresponding week.
Time Frame: Randomization to Last Study Visit (up to 16 weeks)
Population: ITT population included all randomized participants who received the Day 1 intravenous infusion (either tanezumab or placebo infusion). Here "overall number of participants analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Median (Full Range); unit: days
Arm/Group | Tanezumab | Naproxen | Placebo
Number analyzed (Participants) | 88 | 87 | 41
days
  Time to >=30% reduction | 8 [2 to 69] | 7 [2 to 39] | 17 [2 to 49]
  Time to >=50% reduction | 18 [2 to 64] | 41 [2 to 61] | 65 [2 to 102]

10. Secondary Outcome: Total Duration of at Least 30% and 50% Reduction From Baseline in Daily Average Low Back Pain Intensity (LBPI) Score
Description: Total duration of response was defined as the total number of days with >=30% or >=50% reduction from baseline in the daily average LBPI score. Daily average low back pain was assessed on an 11-point numeric rating scale (NRS). Participants described their average low back pain during the past 24 hours on a scale ranging from 0 (no pain) to 10 (worst possible pain), with lower scores indicating less pain. Baseline value was calculated as mean of the scores over 5-day prior to randomization (initial pain assessment period). Post-baseline weekly scores were calculated based on the mean of the scores over the 7 days prior to and including the day at the end of the corresponding week.
Time Frame: Week 1 up to Week 12
Population: ITT population included all randomized participants who received the Day 1 intravenous infusion (either tanezumab or placebo infusion).
Measure: Least Squares Mean (Standard Error); unit: days
Arm/Group | Tanezumab | Naproxen | Placebo
Number analyzed (Participants) | 88 | 88 | 41
days
  Total duration for >=30% reduction | 43.91 (3.54) | 38.81 (3.59) | 33.13 (4.82)
  Total duration for >=50% reduction | 33.21 (3.30) | 27.58 (3.34) | 22.08 (4.49)

11. Secondary Outcome: Change From Baseline in Roland-Morris Disability Questionnaire Total Score at Week 1, 2, 4, 6, 8, and 12
Description: Roland-Morris Disability Questionnaire: low back pain-specific, participant administered questionnaire that assessed how well participants with low back pain were able to function with regard to daily activities. The questionnaire consisted of 24 statements and the participants were instructed to put a mark next to each appropriate statement if it described their pain on the day of assessment. The number of statements marked were added up by the clinician. Total RMDQ score was calculated as the sum of number of statements checked. Total possible score ranged from 0 to 24, with higher scores indicated greater disability.
Time Frame: Baseline, Week 1, 2, 4, 6, 8, 12
Population: ITT population. Here "overall number of participants analyzed" signifies those participants who were evaluable for this outcome measure and 'number analyzed' signifies those participants who were evaluable for this measure at given time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab | Naproxen | Placebo
Number analyzed (Participants) | 87 | 88 | 41
units on a scale
  Baseline | 12.33 (4.63) | 12.36 (4.80) | 13.68 (5.17)
  Change at Week 1: number analyzed (Participants) | 77 | 84 | 41
  Change at Week 1 | -5.21 (5.24) | -3.69 (5.11) | -3.76 (5.25)
  Change at Week 2: number analyzed (Participants) | 76 | 82 | 36
  Change at Week 2 | -5.17 (5.59) | -4.04 (5.37) | -4.08 (6.25)
  Change at Week 4: number analyzed (Participants) | 67 | 79 | 36
  Change at Week 4 | -7.24 (5.33) | -4.00 (4.99) | -4.31 (5.81)
  Change at Week 6: number analyzed (Participants) | 65 | 75 | 31
  Change at Week 6 | -7.88 (5.39) | -4.69 (5.34) | -4.55 (6.55)
  Change at Week 8: number analyzed (Participants) | 60 | 71 | 30
  Change at Week 8 | -7.93 (4.97) | -5.17 (5.32) | -5.60 (6.22)
  Change at Week 12: number analyzed (Participants) | 59 | 67 | 24
  Change at Week 12 | -7.12 (6.00) | -5.10 (5.50) | -4.67 (6.84)

12. Secondary Outcome: Change From Baseline in Modified Brief Pain Inventory-short Form (mBPI-sf) Scores for Pain Interference With Function (Composite Score), General Activity, Walking Ability, Normal Work and Sleep Scores at Week 1, 2, 4, 6, 8 and 12
Description: The mBPI-sf was a self-administered questionnaire used to assess the severity of pain and the impact of pain on daily functions during the 24-hour period prior to evaluation. It consisted of 5 questions. Questions 1 to 4 assessed the magnitude of pain (worst, least, average, right now) on an 11-point NRS ranging from 0 (no pain) to 10 (pain as bad as you can imagine). Question 5 consisted of 7 sub-items (general activity [GA], mood, walking ability [WA], normal work [NW], relations with other people, sleep, enjoyment of life) which measured the level of interference of pain on daily functions. Each sub-item was assessed on an 11-point NRS ranging from 0 (did not interfere) to 10 (completely interfere). The response from 7 sub-items of question 5 were averaged to obtain pain interference composite score (CS), range: 0 to 10 (higher score=more interference).
Time Frame: Baseline, Week 1, 2, 4, 6, 8, 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab | Naproxen | Placebo
Number analyzed (Participants) | 88 | 88 | 41
units on a scale
  Baseline: CS: number analyzed (Participants) | 87 | 88 | 41
  Baseline: CS | 4.81 (2.19) | 5.43 (2.14) | 5.29 (2.25)
  Baseline: GA | 5.55 (2.26) | 5.83 (2.25) | 5.49 (2.72)
  Baseline: WA: number analyzed (Participants) | 87 | 88 | 41
  Baseline: WA | 4.46 (2.80) | 5.25 (2.66) | 5.15 (2.81)
  Baseline: NW: number analyzed (Participants) | 87 | 88 | 41
  Baseline: NW | 5.15 (2.48) | 5.89 (2.38) | 5.80 (2.39)
  Baseline: Sleep: number analyzed (Participants) | 87 | 88 | 41
  Baseline: Sleep | 5.69 (2.70) | 5.75 (2.69) | 6.20 (2.44)
  Change at Week 1: CS: number analyzed (Participants) | 77 | 83 | 41
  Change at Week 1: CS | -2.52 (2.13) | -2.51 (2.46) | -2.07 (2.17)
  Change at Week 1: GA: number analyzed (Participants) | 78 | 83 | 41
  Change at Week 1: GA | -3.10 (2.63) | -2.51 (2.82) | -1.88 (2.47)
  Change at Week 1: WA: number analyzed (Participants) | 77 | 83 | 41
  Change at Week 1: WA | -2.35 (2.64) | -2.04 (2.96) | -2.17 (2.94)
  Change at Week 1: NW: number analyzed (Participants) | 77 | 83 | 41
  Change at Week 1: NW | -2.75 (2.41) | -2.40 (2.84) | -2.22 (2.75)
  Change at Week 1: Sleep: number analyzed (Participants) | 77 | 83 | 41
  Change at Week 1: Sleep | -2.73 (2.52) | -2.87 (3.02) | -2.27 (2.53)
  Change at Week 2: CS: number analyzed (Participants) | 76 | 82 | 36
  Change at Week 2: CS | -2.17 (2.13) | -2.82 (2.41) | -2.70 (2.71)
  Change at Week 2: GA: number analyzed (Participants) | 77 | 82 | 36
  Change at Week 2: GA | -2.61 (2.58) | -2.94 (2.84) | -2.58 (3.54)
  Change at Week 2: WA: number analyzed (Participants) | 76 | 82 | 36
  Change at Week 2: WA | -1.87 (2.94) | -2.48 (2.79) | -2.64 (3.16)
  Change at Week 2: NW: number analyzed (Participants) | 76 | 82 | 36
  Change at Week 2: NW | -2.45 (2.55) | -3.02 (2.61) | -2.92 (3.08)
  Change at Week 2: Sleep: number analyzed (Participants) | 76 | 82 | 36
  Change at Week 2: Sleep | -2.41 (2.49) | -2.88 (2.70) | -3.19 (2.88)
  Change at Week 4: CS: number analyzed (Participants) | 67 | 79 | 36
  Change at Week 4: CS | -3.13 (2.01) | -2.52 (2.35) | -2.72 (2.80)
  Change at Week 4: GA: number analyzed (Participants) | 67 | 79 | 36
  Change at Week 4: GA | -3.62 (2.29) | -2.58 (2.72) | -2.36 (3.87)
  Change at Week 4: WA: number analyzed (Participants) | 68 | 79 | 36
  Change at Week 4: WA | -2.87 (2.50) | -2.09 (2.72) | -2.81 (3.04)
  Change at Week 4: NW: number analyzed (Participants) | 67 | 79 | 36
  Change at Week 4: NW | -3.55 (2.36) | -2.63 (2.65) | -2.81 (3.25)
  Change at Week 4: Sleep: number analyzed (Participants) | 67 | 79 | 36
  Change at Week 4: Sleep | -3.54 (2.51) | -2.63 (3.20) | -3.08 (2.90)
  Change at Week 6: CS: number analyzed (Participants) | 65 | 75 | 31
  Change at Week 6: CS | -3.25 (1.85) | -2.84 (2.29) | -2.76 (2.61)
  Change at Week 6: GA: number analyzed (Participants) | 66 | 75 | 31
  Change at Week 6: GA | -3.65 (2.12) | -2.97 (2.66) | -2.68 (3.07)
  Change at Week 6: WA: number analyzed (Participants) | 65 | 75 | 31
  Change at Week 6: WA | -3.11 (2.55) | -2.48 (2.86) | -2.39 (2.84)
  Change at Week 6: NW: number analyzed (Participants) | 65 | 75 | 31
  Change at Week 6: NW | -3.55 (2.04) | -2.95 (2.74) | -2.87 (3.12)
  Change at Week 6: Sleep: number analyzed (Participants) | 65 | 75 | 31
  Change at Week 6: Sleep | -3.92 (2.54) | -2.99 (2.95) | -3.03 (2.58)
  Change at Week 8: CS: number analyzed (Participants) | 60 | 71 | 30
  Change at Week 8: CS | -3.19 (1.84) | -3.01 (2.31) | -3.04 (2.73)
  Change at Week 8: GA: number analyzed (Participants) | 61 | 71 | 30
  Change at Week 8: GA | -3.72 (2.22) | -3.14 (2.78) | -2.93 (3.27)
  Change at Week 8: WA: number analyzed (Participants) | 60 | 71 | 30
  Change at Week 8: WA | -3.05 (2.56) | -2.62 (3.04) | -2.87 (3.07)
  Change at Week 8: NW: number analyzed (Participants) | 60 | 71 | 30
  Change at Week 8: NW | -3.62 (2.08) | -3.24 (2.59) | -3.33 (3.13)
  Change at Week 8: Sleep: number analyzed (Participants) | 60 | 71 | 30
  Change at Week 8: Sleep | -3.47 (2.45) | -3.51 (2.93) | -3.33 (2.80)
  Change at Week 12: CS: number analyzed (Participants) | 59 | 67 | 24
  Change at Week 12: CS | -3.08 (2.01) | -2.84 (2.34) | -2.74 (3.15)
  Change at Week 12: GA: number analyzed (Participants) | 60 | 67 | 24
  Change at Week 12: GA | -3.45 (2.42) | -3.01 (2.93) | -2.92 (3.79)
  Change at Week 12: WA: number analyzed (Participants) | 59 | 67 | 24
  Change at Week 12: WA | -2.78 (2.71) | -2.54 (2.87) | -2.04 (3.48)
  Change at Week 12: NW: number analyzed (Participants) | 59 | 67 | 24
  Change at Week 12: NW | -3.36 (2.43) | -2.97 (2.63) | -3.17 (3.29)
  Change at Week 12: Sleep: number analyzed (Participants) | 59 | 67 | 24
  Change at Week 12: Sleep | -3.58 (2.44) | -3.33 (2.87) | -3.08 (2.80)

13. Secondary Outcome: Number of Participants With Change From Baseline in Patient's Global Assessment of Low Back Pain (Disease Activity) Score at Week 1, 2, 4, 6, 8 and 12
Description: Patient's global assessment of low back pain scale assessed participants overall impression of disease activity. Participants answered: "Considering all the ways your low back pain affects you, how are you doing today?" Participants responded using a 5-point Likert scale with a score of 1 being the best (very good) and a score of 5 being the worst (very poor). Participants who reported a change of -4, -3, -2, -1, 0, 1, 2, 3, 4 from Baseline in Patient's Global Assessment of Low Back Pain (Disease Activity) score at specified weeks were presented.
Time Frame: Week 1, 2, 4, 6, 8, 12
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab | Naproxen | Placebo
Number analyzed (Participants) | 77 | 84 | 41
Participants
  Week 1: Change= -4 | 1 | 0 | 0
  Week 1: Change= -3 | 1 | 2 | 1
  Week 1: Change= -2 | 24 | 18 | 6
  Week 1: Change= -1 | 23 | 33 | 14
  Week 1: Change= 0 | 25 | 26 | 17
  Week 1: Change= 1 | 2 | 4 | 3
  Week 1: Change= 2 | 1 | 1 | 0
  Week 1: Change= 3 | 0 | 0 | 0
  Week 1: Change= 4 | 0 | 0 | 0
  Week 2: Change= -4: number analyzed (Participants) | 76 | 82 | 36
  Week 2: Change= -4 | 1 | 1 | 0
  Week 2: Change= -3: number analyzed (Participants) | 76 | 82 | 36
  Week 2: Change= -3 | 2 | 4 | 4
  Week 2: Change= -2: number analyzed (Participants) | 76 | 82 | 36
  Week 2: Change= -2 | 16 | 17 | 5
  Week 2: Change= -1: number analyzed (Participants) | 76 | 82 | 36
  Week 2: Change= -1 | 26 | 30 | 17
  Week 2: Change= 0: number analyzed (Participants) | 76 | 82 | 36
  Week 2: Change= 0 | 24 | 23 | 8
  Week 2: Change= 1: number analyzed (Participants) | 76 | 82 | 36
  Week 2: Change= 1 | 6 | 6 | 2
  Week 2: Change= 2: number analyzed (Participants) | 76 | 82 | 36
  Week 2: Change= 2 | 1 | 1 | 0
  Week 2: Change= 3: number analyzed (Participants) | 76 | 82 | 36
  Week 2: Change= 3 | 0 | 0 | 0
  Week 2: Change= 4: number analyzed (Participants) | 76 | 82 | 36
  Week 2: Change= 4 | 0 | 0 | 0
  Week 4: Change= -4: number analyzed (Participants) | 67 | 79 | 36
  Week 4: Change= -4 | 1 | 1 | 0
  Week 4: Change= -3: number analyzed (Participants) | 67 | 79 | 36
  Week 4: Change= -3 | 0 | 2 | 5
  Week 4: Change= -2: number analyzed (Participants) | 67 | 79 | 36
  Week 4: Change= -2 | 22 | 18 | 6
  Week 4: Change= -1: number analyzed (Participants) | 67 | 79 | 36
  Week 4: Change= -1 | 30 | 32 | 15
  Week 4: Change= 0: number analyzed (Participants) | 67 | 79 | 36
  Week 4: Change= 0 | 14 | 20 | 7
  Week 4: Change= 1: number analyzed (Participants) | 67 | 79 | 36
  Week 4: Change= 1 | 0 | 4 | 3
  Week 4: Change= 2: number analyzed (Participants) | 67 | 79 | 36
  Week 4: Change= 2 | 0 | 2 | 0
  Week 4: Change= 3: number analyzed (Participants) | 67 | 79 | 36
  Week 4: Change= 3 | 0 | 0 | 0
  Week 4: Change= 4: number analyzed (Participants) | 67 | 79 | 36
  Week 4: Change= 4 | 0 | 0 | 0
  Week 6: Change= -4: number analyzed (Participants) | 65 | 75 | 31
  Week 6: Change= -4 | 2 | 0 | 0
  Week 6: Change= -3: number analyzed (Participants) | 65 | 75 | 31
  Week 6: Change= -3 | 2 | 7 | 3
  Week 6: Change= -2: number analyzed (Participants) | 65 | 75 | 31
  Week 6: Change= -2 | 25 | 22 | 5
  Week 6: Change= -1: number analyzed (Participants) | 65 | 75 | 31
  Week 6: Change= -1 | 20 | 18 | 12
  Week 6: Change= 0: number analyzed (Participants) | 65 | 75 | 31
  Week 6: Change= 0 | 15 | 20 | 10
  Week 6: Change= 1: number analyzed (Participants) | 65 | 75 | 31
  Week 6: Change= 1 | 1 | 7 | 1
  Week 6: Change= 2: number analyzed (Participants) | 65 | 75 | 31
  Week 6: Change= 2 | 0 | 1 | 0
  Week 6: Change= 3: number analyzed (Participants) | 65 | 75 | 31
  Week 6: Change= 3 | 0 | 0 | 0
  Week 6: Change= 4: number analyzed (Participants) | 65 | 75 | 31
  Week 6: Change= 4 | 0 | 0 | 0
  Week 8: Change= -4: number analyzed (Participants) | 60 | 71 | 30
  Week 8: Change= -4 | 0 | 0 | 0
  Week 8: Change= -3: number analyzed (Participants) | 60 | 71 | 30
  Week 8: Change= -3 | 2 | 5 | 2
  Week 8: Change= -2: number analyzed (Participants) | 60 | 71 | 30
  Week 8: Change= -2 | 23 | 17 | 6
  Week 8: Change= -1: number analyzed (Participants) | 60 | 71 | 30
  Week 8: Change= -1 | 23 | 25 | 14
  Week 8: Change= 0: number analyzed (Participants) | 60 | 71 | 30
  Week 8: Change= 0 | 11 | 19 | 4
  Week 8: Change= 1: number analyzed (Participants) | 60 | 71 | 30
  Week 8: Change= 1 | 1 | 4 | 4
  Week 8: Change= 2: number analyzed (Participants) | 60 | 71 | 30
  Week 8: Change= 2 | 0 | 1 | 0
  Week 8: Change= 3: number analyzed (Participants) | 60 | 71 | 30
  Week 8: Change= 3 | 0 | 0 | 0
  Week 8: Change= 4: number analyzed (Participants) | 60 | 71 | 30
  Week 8: Change= 4 | 0 | 0 | 0
  Week 12: Change= -4: number analyzed (Participants) | 59 | 67 | 24
  Week 12: Change= -4 | 1 | 0 | 0
  Week 12: Change= -3: number analyzed (Participants) | 59 | 67 | 24
  Week 12: Change= -3 | 1 | 6 | 4
  Week 12: Change= -2: number analyzed (Participants) | 59 | 67 | 24
  Week 12: Change= -2 | 14 | 15 | 2
  Week 12: Change= -1: number analyzed (Participants) | 59 | 67 | 24
  Week 12: Change= -1 | 22 | 21 | 9
  Week 12: Change= 0: number analyzed (Participants) | 59 | 67 | 24
  Week 12: Change= 0 | 20 | 14 | 7
  Week 12: Change= 1: number analyzed (Participants) | 59 | 67 | 24
  Week 12: Change= 1 | 1 | 11 | 1
  Week 12: Change= 2: number analyzed (Participants) | 59 | 67 | 24
  Week 12: Change= 2 | 0 | 0 | 1
  Week 12: Change= 3: number analyzed (Participants) | 59 | 67 | 24
  Week 12: Change= 3 | 0 | 0 | 0
  Week 12: Change= 4: number analyzed (Participants) | 59 | 67 | 24
  Week 12: Change= 4 | 0 | 0 | 0

14. Secondary Outcome: Number of Participants With Each Response Level of Patient's Global Evaluation of Study Medication
Description: Participants answered: "In all ways, how would you rate your overall response to the study medication today?" Participants responded using a 4-point Likert scale where 1 = poor, 2 = fair, 3 = good and 4 = excellent. Higher score indicated better overall response to the treatment.
Time Frame: Week 1, 2, 4, 6, 8, 12
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab | Naproxen | Placebo
Number analyzed (Participants) | 78 | 84 | 40
Participants
  Week 1: Poor | 7 | 13 | 12
  Week 1: Fair | 16 | 22 | 11
  Week 1: Good | 29 | 32 | 14
  Week 1: Excellent | 26 | 17 | 3
  Week 2: Poor: number analyzed (Participants) | 77 | 82 | 36
  Week 2: Poor | 10 | 16 | 6
  Week 2: Fair: number analyzed (Participants) | 77 | 82 | 36
  Week 2: Fair | 17 | 14 | 11
  Week 2: Good: number analyzed (Participants) | 77 | 82 | 36
  Week 2: Good | 31 | 34 | 15
  Week 2: Excellent: number analyzed (Participants) | 77 | 82 | 36
  Week 2: Excellent | 19 | 18 | 4
  Week 4: Poor: number analyzed (Participants) | 68 | 79 | 36
  Week 4: Poor | 4 | 15 | 8
  Week 4: Fair: number analyzed (Participants) | 68 | 79 | 36
  Week 4: Fair | 5 | 16 | 10
  Week 4: Good: number analyzed (Participants) | 68 | 79 | 36
  Week 4: Good | 30 | 27 | 13
  Week 4: Excellent: number analyzed (Participants) | 68 | 79 | 36
  Week 4: Excellent | 29 | 21 | 5
  Week 6: Poor: number analyzed (Participants) | 65 | 75 | 31
  Week 6: Poor | 1 | 11 | 8
  Week 6: Fair: number analyzed (Participants) | 65 | 75 | 31
  Week 6: Fair | 10 | 23 | 5
  Week 6: Good: number analyzed (Participants) | 65 | 75 | 31
  Week 6: Good | 22 | 23 | 14
  Week 6: Excellent: number analyzed (Participants) | 65 | 75 | 31
  Week 6: Excellent | 32 | 18 | 4
  Week 8: Poor: number analyzed (Participants) | 61 | 71 | 30
  Week 8: Poor | 1 | 9 | 6
  Week 8: Fair: number analyzed (Participants) | 61 | 71 | 30
  Week 8: Fair | 8 | 24 | 7
  Week 8: Good: number analyzed (Participants) | 61 | 71 | 30
  Week 8: Good | 20 | 19 | 13
  Week 8: Excellent: number analyzed (Participants) | 61 | 71 | 30
  Week 8: Excellent | 32 | 19 | 4
  Week 12: Poor: number analyzed (Participants) | 59 | 67 | 24
  Week 12: Poor | 6 | 15 | 6
  Week 12: Fair: number analyzed (Participants) | 59 | 67 | 24
  Week 12: Fair | 9 | 17 | 6
  Week 12: Good: number analyzed (Participants) | 59 | 67 | 24
  Week 12: Good | 21 | 18 | 5
  Week 12: Excellent: number analyzed (Participants) | 59 | 67 | 24
  Week 12: Excellent | 23 | 17 | 7

15. Secondary Outcome: Number of Participants Who Discontinued the Study Due to Lack of Efficacy
Time Frame: Baseline up to Week 12
Population: Safety population included all randomized participants who received the Day 1 intravenous infusion (either tanezumab or placebo infusion).
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab | Naproxen | Placebo
Number analyzed (Participants) | 88 | 88 | 41
Participants | 7 | 14 | 8

16. Secondary Outcome: Time to Discontinuation Due to Lack of Efficacy
Description: Median time to discontinuation due to lack of efficacy was estimated using Kaplan-Meier method. Median was not estimable if the percentage of participants who discontinued due to lack of efficacy was below 50%.
Time Frame: Baseline up to Week 12
Population: as for outcome 15
Measure: Median (Full Range); unit: days
Arm/Group | Tanezumab | Naproxen | Placebo
Number analyzed (Participants) | 88 | 88 | 41
days | NA [8 to 49] — Median was not evaluable since very low number of participants discontinued due to lack of efficacy. | NA [9 to 71] — Median was not evaluable since very low number of participants discontinued due to lack of efficacy. | NA [6 to 57] — Median was not evaluable since very low number of participants discontinued due to lack of efficacy.

17. Secondary Outcome: Number of Participants With Chronic Low Back Pain (CLBP) Response
Description: Participants were considered as CLBP responders if they had achieved a reduction of >=30% in daily average LBPI score from baseline, an increase of >=30% in patient's global assessment of low back pain (disease activity) from baseline, and no worsening (increase) in RMDQ total score from baseline at specified week. Daily average low back pain assessed on an 11-point NRS ranging from 0 (no pain) to 10 (worst possible pain). Patient's global assessment of low back pain assessed using a 5-point Likert scale with a score of 1 being the best (very good) and a score of 5 being the worst (very poor). RMDQ: low back pain-specific, participant administered questionnaire consisted of 24 statements and participants were instructed to put a mark next to each appropriate statement if it described their pain on the day of assessment. Total RMDQ score was calculated as sum of number of statements checked. Total possible score ranged from 0 to 24, with higher scores indicated greater disability.
Time Frame: Weeks 1, 2, 4, 6, 8, 12
Population: ITT population included all randomized participants who received the Day 1 intravenous infusion (either tanezumab or placebo infusion). LOCF method was used to impute missing values. Here "overall number of participants analyzed" signifies those participants who were evaluable for this outcome measure
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab | Naproxen | Placebo
Number analyzed (Participants) | 87 | 88 | 41
Participants
  Week 1 | 33 | 30 | 6
  Week 2 | 32 | 34 | 9
  Week 4 | 51 | 31 | 11
  Week 6 | 50 | 39 | 9
  Week 8 | 48 | 36 | 14
  Week 12 | 38 | 30 | 12

18. Secondary Outcome: Number of Participants Who Used Rescue Medications
Description: In case of inadequate pain relief for CLBP or for non-CLBP related pain, acetaminophen up to 2000 mg per day up to 3 days per week could be taken as rescue medication. Number of participants with any use of rescue medication during the particular study week were summarized.
Time Frame: Week 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12
Population: Safety population included all randomized participants who received the Day 1 intravenous infusion (either tanezumab or placebo infusion). Here 'number analyzed' signifies those participants who were evaluable for this measure at given time points.
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab | Naproxen | Placebo
Number analyzed (Participants) | 88 | 88 | 41
Participants
  Week 1 | 61 | 50 | 29
  Week 2: number analyzed (Participants) | 88 | 87 | 40
  Week 2 | 65 | 49 | 27
  Week 3: number analyzed (Participants) | 81 | 84 | 38
  Week 3 | 54 | 42 | 24
  Week 4: number analyzed (Participants) | 77 | 80 | 38
  Week 4 | 40 | 49 | 28
  Week 5: number analyzed (Participants) | 75 | 80 | 36
  Week 5 | 37 | 46 | 21
  Week 6: number analyzed (Participants) | 72 | 77 | 34
  Week 6 | 36 | 42 | 20
  Week 7: number analyzed (Participants) | 72 | 75 | 33
  Week 7 | 34 | 38 | 17
  Week 8: number analyzed (Participants) | 67 | 73 | 33
  Week 8 | 31 | 39 | 19
  Week 9: number analyzed (Participants) | 66 | 72 | 32
  Week 9 | 33 | 38 | 12
  Week 10: number analyzed (Participants) | 64 | 72 | 29
  Week 10 | 30 | 41 | 14
  Week 11: number analyzed (Participants) | 64 | 72 | 28
  Week 11 | 32 | 31 | 13
  Week 12: number analyzed (Participants) | 64 | 71 | 27
  Week 12 | 30 | 33 | 16

19. Secondary Outcome: Duration of Rescue Medication Use
Description: In case of inadequate pain relief for CLBP or for non-CLBP related pain, acetaminophen up to 2000 mg per day up to 3 days per week could be taken as rescue medication. The number of days of rescue medication use during the particular week were summarized.
Time Frame: Week 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12
Population: as for outcome 18
Measure: Median (Full Range); unit: days
Arm/Group | Tanezumab | Naproxen | Placebo
Number analyzed (Participants) | 88 | 88 | 41
days
  Week 1 | 2 [0 to 6] | 1 [0 to 6] | 1 [0 to 6]
  Week 2: number analyzed (Participants) | 88 | 87 | 40
  Week 2 | 2 [0 to 7] | 1 [0 to 7] | 1.5 [0 to 7]
  Week 3: number analyzed (Participants) | 81 | 84 | 38
  Week 3 | 2 [0 to 7] | 0.5 [0 to 7] | 2 [0 to 7]
  Week 4: number analyzed (Participants) | 77 | 80 | 38
  Week 4 | 1 [0 to 7] | 2 [0 to 7] | 2 [0 to 7]
  Week 5: number analyzed (Participants) | 75 | 80 | 36
  Week 5 | 0 [0 to 7] | 1 [0 to 7] | 1 [0 to 7]
  Week 6: number analyzed (Participants) | 72 | 77 | 34
  Week 6 | 0.5 [0 to 7] | 1 [0 to 7] | 1 [0 to 7]
  Week 7: number analyzed (Participants) | 72 | 75 | 33
  Week 7 | 0 [0 to 7] | 1 [0 to 7] | 1 [0 to 7]
  Week 8: number analyzed (Participants) | 67 | 73 | 33
  Week 8 | 0 [0 to 7] | 1 [0 to 7] | 1 [0 to 7]
  Week 9: number analyzed (Participants) | 66 | 72 | 32
  Week 9 | 0.5 [0 to 7] | 1 [0 to 7] | 0 [0 to 7]
  Week 10: number analyzed (Participants) | 64 | 72 | 29
  Week 10 | 0 [0 to 7] | 1 [0 to 7] | 0 [0 to 7]
  Week 11: number analyzed (Participants) | 64 | 72 | 28
  Week 11 | 0.5 [0 to 7] | 0 [0 to 7] | 0 [0 to 7]
  Week 12: number analyzed (Participants) | 64 | 71 | 27
  Week 12 | 0 [0 to 7] | 0 [0 to 7] | 1 [0 to 7]

20. Secondary Outcome: Amount of Rescue Medication Taken
Description: In case of inadequate pain relief for CLBP or for non-CLBP related pain, acetaminophen up to 2000 mg per day up to 3 days per week could be taken as rescue medication. The total dosage of acetaminophen (in mg) in each particular week was summarized.
Time Frame: Week 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Tanezumab | Naproxen | Placebo
Number analyzed (Participants) | 88 | 88 | 41
mg
  Week 1 | 2545.5 (2798.4) | 2039.8 (2467.3) | 2451.2 (2816.9)
  Week 2: number analyzed (Participants) | 88 | 87 | 40
  Week 2 | 3221.6 (3528.1) | 2327.6 (3083.0) | 2225.0 (2616.4)
  Week 3: number analyzed (Participants) | 81 | 84 | 38
  Week 3 | 2703.7 (3368.8) | 2208.3 (3112.6) | 2565.8 (2719.2)
  Week 4: number analyzed (Participants) | 77 | 80 | 38
  Week 4 | 2220.8 (3108.2) | 2475.0 (2937.0) | 2434.2 (2904.3)
  Week 5: number analyzed (Participants) | 75 | 80 | 36
  Week 5 | 2073.3 (3100.5) | 2318.8 (2936.3) | 2444.4 (3285.9)
  Week 6: number analyzed (Participants) | 72 | 77 | 34
  Week 6 | 2062.5 (2919.0) | 2227.3 (3193.9) | 2573.5 (3348.7)
  Week 7: number analyzed (Participants) | 72 | 75 | 33
  Week 7 | 1854.2 (3126.9) | 1873.3 (2763.3) | 2393.9 (3149.3)
  Week 8: number analyzed (Participants) | 67 | 73 | 33
  Week 8 | 2134.3 (3273.6) | 2212.3 (3255.2) | 1924.2 (2478.4)
  Week 9: number analyzed (Participants) | 66 | 72 | 32
  Week 9 | 1772.7 (2627.1) | 2319.4 (3483.7) | 1406.3 (2554.1)
  Week 10: number analyzed (Participants) | 64 | 72 | 29
  Week 10 | 1851.6 (2655.8) | 2513.9 (3477.3) | 1534.5 (2591.0)
  Week 11: number analyzed (Participants) | 64 | 72 | 28
  Week 11 | 1992.2 (2717.5) | 2166.7 (3632.8) | 1375.0 (2311.9)
  Week 12: number analyzed (Participants) | 64 | 71 | 27
  Week 12 | 1828.1 (2790.6) | 2253.5 (3402.6) | 1722.2 (2805.7)

21. Other Pre Specified Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) or Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 28 days after last dose (up to Week 16) that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: Baseline up to 28 days after last dose of study treatment (up to Week 16)
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab | Naproxen | Placebo
Number analyzed (Participants) | 88 | 88 | 41
Participants
  AEs | 50 | 54 | 27
  SAEs | 0 | 2 | 0

22. Other Pre Specified Outcome: Number of Participants With Anti-Drug Antibody (ADA)
Description: Human serum anti-drug antibody (ADA) samples were analyzed for the presence or absence of anti-tanezumab antibodies by using the semi-quantitative enzyme-linked immunosorbent assay (ELISA).
Time Frame: Baseline up to Week 12
Population: Safety population included all randomized participants who received the Day 1 intravenous infusion of tanezumab. Data for this outcome measure was not planned to be collected and analyzed for Naproxen and Placebo arms.
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab
Number analyzed (Participants) | 88
Participants | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Tanezumab | Naproxen | Placebo
Serious Adverse Events (participants affected / at risk) | 0/88 | 2/88 | 0/41
Other Adverse Events (participants affected / at risk) | 44/88 | 45/88 | 27/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tanezumab (N=88) | Naproxen (N=88) | Placebo (N=41)
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0
Syncope vasovagal (Nervous system disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tanezumab (N=88) | Naproxen (N=88) | Placebo (N=41)
Vertigo (Ear and labyrinth disorders) | 2 | 1 | 0
Conjunctivitis (Eye disorders) | 2 | 0 | 0
Diplopia (Eye disorders) | 0 | 0 | 1
Dry eye (Eye disorders) | 0 | 0 | 1
Vision blurred (Eye disorders) | 2 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 4 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 3
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 2 | 0
Nausea (Gastrointestinal disorders) | 2 | 1 | 1
Stomach discomfort (Gastrointestinal disorders) | 0 | 1 | 1
Chest discomfort (General disorders) | 2 | 0 | 0
Chest pain (General disorders) | 1 | 1 | 1
Fatigue (General disorders) | 2 | 1 | 1
Influenza like illness (General disorders) | 1 | 0 | 1
Seasonal allergy (Immune system disorders) | 0 | 2 | 1
Bronchitis (Infections and infestations) | 2 | 0 | 2
Ear infection (Infections and infestations) | 3 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 1
Influenza (Infections and infestations) | 3 | 5 | 1
Nasopharyngitis (Infections and infestations) | 2 | 6 | 1
Sinusitis (Infections and infestations) | 1 | 5 | 0
Upper respiratory tract infection (Infections and infestations) | 4 | 4 | 2
Urinary tract infection (Infections and infestations) | 3 | 4 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 6 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 2
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Joint sprain (Injury, poisoning and procedural complications) | 3 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 2 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 | 6 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 5 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 7 | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 2 | 2
Dysaesthesia (Nervous system disorders) | 2 | 0 | 0
Headache (Nervous system disorders) | 10 | 5 | 8
Hyperaesthesia (Nervous system disorders) | 6 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1
Pallanaesthesia (Nervous system disorders) | 0 | 2 | 0
Paraesthesia (Nervous system disorders) | 4 | 1 | 0
Restless legs syndrome (Nervous system disorders) | 0 | 0 | 1
Sinus headache (Nervous system disorders) | 2 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 1
Abnormal dreams (Psychiatric disorders) | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 2 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Flushing (Vascular disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.